CLINICAL TRIAL: NCT06020300
Title: Short Course Low Dose Oral Colchicine After ST Elevation Myocardial Infarction(STEMI)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FF-2023-191
Record Dates: First submitted 2023-08-03; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Colchicine; Tablets; Pyridoxine

STUDY DESIGN:
Intervention Model Description: Block randomization method will be used for sampling. Patients recruited will be randomly assigned to colchicine & placebo group with 1:1 ratio
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Tablet Pyridoxine used as placebo in view of tablet colchicine look alike
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine Post ST Elevation Myocardial Infarction (STEMI) (Experimental): 32 patients with STEMI are assigned for oral colchicine 0.6 mg once daily upon admission for 30 days
  Interventions: Drug: Oral Colchicine 0.6 mg
- Placebo (Pyridoxine) Post ST Elevation myocardial Infraction (STEMI) (Placebo Comparator): Another 32 patients with STEMI are assigned for placebo (oral pyridoxine 10 mg) once daily upon admission for 30 days
  Interventions: Drug: Oral Pyridoxine 10 mg

INTERVENTIONS:
Drug: Oral Colchicine 0.6 mg — Anti-Inflammatory Effects
  Other Names: GOUTNOR 0.6 mg Tablet
  Arms: Colchicine Post ST Elevation Myocardial Infarction (STEMI)
Drug: Oral Pyridoxine 10 mg — Colchicine look alike placebo
  Other Names: MSA Pyridoxine HCI 10 mg Tablet
  Arms: Placebo (Pyridoxine) Post ST Elevation myocardial Infraction (STEMI)

SUMMARY:
To Study Efficacy and safety oral colchicine 0.6 mg post ST Elevation myocardial infraction (STEMI)

DETAILED DESCRIPTION:
Colchicine is a cheap and potent anti-inflammatory. We believe anti-inflammatory is able to reduce inflammation in coronary arteries and heart muscle post ST elevation myocardial infarction which may benefit in short and long term outcome in patients. The short term outcome is measured using serum troponin and long term outcome is assessed with transthoracic echocardiogram and major adverse cardiac events.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 years to 80 years old
2. STEMI within 24 hours of admission to Pusat Perubatan UKM & undergoing revascularization therapy (percutaneous coronary intervention) during admission

STEMI is diagnosed when there is:

* ST elevation of ≥1 mm in 2 contiguous leads or
* a new onset LBBB in the resting ECG
* in a patient with ischaemic type chest pains of > 30 minutes and
* accompanied by a rise and fall in cardiac biomarkers (CPG MALAYSIA STEMI 2019, 4th Edition)

Exclusion Criteria:

1. Pre-existing severe heart failure with left ventricular ejection fraction less than 35%
2. Clinically unstable (Intubated or double inotropic support)
3. Refuse or not suitable for cardiac revascularization therapy
4. Anaemia induced Angina (Hb < 9 g/dL)
5. Ongoing sepsis requiring antibiotic
6. Ongoing diarrhea (Loose stool 3 times or more per day - stool consistency Bristol chart type 6 & 7)
7. Active Covid-19 Infection (< 7 days for Category 1-3, < 10 days for category 4-5)
8. Stroke within previous 3 months
9. Coronary bypass surgery either within the previous 3 years or planned
10. Active malignancy or treated malignancy within 7 years
11. Active Inflammatory bowel disease on treatment
12. Active Neuromuscular disease on treatment
13. Chronic kidney disease (CKD stage 4 - eGFR < 30 mL/min/1.73 m2)
14. Severe hepatic disease (ALT > 3X upper limit normal, Bilirubin > 2X upper limit normal)
15. Active drug or alcohol abuse on therapy
16. On long term or recent systemic glucocorticoid therapy within 3 months
17. Pregnancy or breastfeeding
18. Known sensitivity to colchicine or multivitamin tablet
19. Pre-existing indication for colchicine therapy (Gout, Familial Mediterranean fever, etc)
20. Patients on oral medications that may interact with colchicine (Clarithromycin, Ketoconazole, Voriconazole, Fluconazole, Itraconazole, Cyclosporine, Ritonavir)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2023-12-29 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Anti-Inflammatory Effect of Colchicine | 3-7 days
  Serum Troponin I change from arrival to discharge
Major Adverse Cardiac Events (MACE) | 3 months
  Recurrent myocardial infarction, unstable angina needing hospital admission, cardiac death, unplanned repeated revascularization, cerebrovascular accident

SECONDARY OUTCOMES:
Trans thoracic Echo cardiogram parameters | 3 months
  Left ventricular ejection fraction (biplane mode) measured in %, left ventricular volume measured in milliliters, left atrial volume measured in milliliters, E/A ratio, E/e ' ratio
Safety of colchicine | 1 month
  Number of Participants with medication side effects

CONTACTS AND LOCATIONS:
Overall Officials: HAMAT HAMDI, MBBchBAO, Principal Investigator — Head of Cardiology Unit
Locations (1):
- Nationa University of Malaysia, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No